CLINICAL TRIAL: NCT03700554
Title: ASPIRATE Study- Comparison of Efficacy and Analgesic Use During the Therapy of Iatrogenic Pneumothorax Using Pleuralvent™ and Large Bore Chest Tube (16F)
Brief Title: Efficacy and Analgesic Use During the Therapy of Iatrogenic Pneumothorax Using Pleuralvent™ and Chest Tube
Acronym: ASPIRATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Olomouc (Other)
Collaborators: Thomayer University Hospital (Other)
Responsible Party: Principal Investigator, Milan Sova, MD, Ph.D., University Hospital Olomouc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASPIRATE
Record Dates: First submitted 2018-10-01; First posted 2018-10-09 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Pneumothorax
Keywords: Pneumothorax; Iatrogenic; Chest tube; Pleuralvent
MeSH Terms: conditions — Pneumothorax | interventions — Chest Tubes

STUDY DESIGN:
Intervention Model Description: Randomised, non-blinded, actively controlled clinical trial.
Who Masked: Investigator
Masking Description: Method of closed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pleuralvent™ (Experimental): Patients treated with Pleuralvent™ device
  Interventions: Device: Pleuralvent™
- Chest tube (Active Comparator): Patients treated with Chest tube
  Interventions: Procedure: Chest tube

INTERVENTIONS:
Device: Pleuralvent™ — Pneumothorax treatment with Pleuralvent™ device (Heimlich valve device)
  Arms: Pleuralvent™
Procedure: Chest tube — Chest tube insertion
  Arms: Chest tube

SUMMARY:
The aim of this clinical trial is to compare the efficiency and analgesic use in the therapy of iatrogenic Pneumothorax when using the Pleuralvent™ system in comparison with large bore chest tubes (catheter 16F).

DETAILED DESCRIPTION:
Rationale:

Pneumothorax is a common, usually invasively treated, disorder. The usual methods of treatment are needle aspiration (14-16 G needles) or chest drainage (16+ F catheters).

A third therapeutic option is the use of small calibre catheters (< 16F). According to some studies, the success rates of these methods are comparable. These catheters have the same success rate as large bore chest tubes and treatment with them is less painful for patients.

The use of Heimlich valves allows for increased patient mobility - or even out-patient treatment.

According to a review by the European Respiratory Society, nowadays there is an availability of systems which are part of advanced intervention techniques. These devices are designed for ease of insertion allowing for the full mobility of patients. It is, however, not clear whether treatment with these new systems is less painful.

The aim of this clinical trial is to compare the efficiency and analgesic use in the therapy of iatrogenic Pneumothorax when using the Pleuralvent™ system in comparison with large bore chest tubes (catheter 16F).

Process:

Following the completion of the initial screening (fulfilling of both inclusion and exclusion criteria) and the signing of informed consent, a patient with iatrogenic pneumothorax (PNO) will be treated with, according to randomisation, either the Pleuralvent™ system or with a large bore chest tube - 16F. A control chest X-ray will be performed immediately after the introduction of the therapeutic method and following 3 days of therapy.

If no signs of PNO are present, the therapy will be terminated. In cases where the lung will not be completely expanded, the control X-ray will be repeated on the 5th, 7th and 10th day of therapy. If, following this, the PNO will persist without resolution, the therapy will be declared non-effective and other therapy modes will be used (conversion to large bore chest drainage in the Pleuralvent™group and surgical treatment in the chest drainage group).

ELIGIBILITY:
Inclusion Criteria:

* Iatrogenic pneumothorax indicated for invasive therapy

Exclusion Criteria:

* Chronic analgesic therapy
* Contraindications for Pleuralvent™ use
* Non-compliance of patients
* Clinically significant hepatopathy (alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 3 times normal values)
* Clinically significant renal insufficiency (glomerular filtration < 0.5 ml/kg/min)
* Allergy to metamizole/tramadol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2019-02-03 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Treatment efficiency | up to 10 days of treatment or until the treatment is terminated
  Condition with no need for further therapy modes defined as a absence of pneumothorax on chest X-ray

SECONDARY OUTCOMES:
Analgesic use | up to 10 days of treatment or until the treatment is terminated
  Comparison of analgesic use in groups - with Pleuralvent™ or large bore chest tube therapy
The time to lung re-expansion | up to 10 days of treatment or until the treatment is terminated
  The treatment duration needed to lung re-expansion
Subjective pain perception according to Visual Analogue Scale (VAS) scale | up to 10 days of treatment or until the treatment is terminated
  Subjective pain perception according to Visual Analogue Scale (scale 0-10, where 0 represents no pain and 10 excruciating pain)

CONTACTS AND LOCATIONS:
Overall Officials: Milan Sova, MD, Ph.D., Principal Investigator — Department of Pulmonary Diseases and Tuberculosis Respiratory Medicine, Faculty of Medicine and Dentistry, Palacky University Olomouc and University Hospital, Olomouc, Czech Republic
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be available upon legitimate request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available after completion of the study
Access Criteria: Upon request

REFERENCES:
- [Background] MacDuff A, Arnold A, Harvey J; BTS Pleural Disease Guideline Group. Management of spontaneous pneumothorax: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii18-31. doi: 10.1136/thx.2010.136986. No abstract available. PMID 20696690
- [Background] Horsley A, Jones L, White J, Henry M. Efficacy and complications of small-bore, wire-guided chest drains. Chest. 2006 Dec;130(6):1857-63. doi: 10.1378/chest.130.6.1857. PMID 17167009
- [Background] Funaki B. Pneumothorax treated by small-bore chest tube. Semin Intervent Radiol. 2007 Jun;24(2):272-6. doi: 10.1055/s-2007-980051. No abstract available. PMID 21326805
- [Background] Vedam H, Barnes DJ. Comparison of large- and small-bore intercostal catheters in the management of spontaneous pneumothorax. Intern Med J. 2003 Nov;33(11):495-9. doi: 10.1046/j.1445-5994.2003.00467.x. PMID 14656251
- [Background] Akowuah E, Ho EC, George R, Brennan K, Tennant S, Braidley P, Cooper G. Less pain with flexible fluted silicone chest drains than with conventional rigid chest tubes after cardiac surgery. J Thorac Cardiovasc Surg. 2002 Nov;124(5):1027-8. doi: 10.1067/mtc.2002.125641. No abstract available. PMID 12407390
- [Background] Bhatnagar R, Corcoran JP, Maldonado F, Feller-Kopman D, Janssen J, Astoul P, Rahman NM. Advanced medical interventions in pleural disease. Eur Respir Rev. 2016 Jun;25(140):199-213. doi: 10.1183/16000617.0020-2016. PMID 27246597
- [Derived] Sova M, Poruba M, Genzor S, Jakubec P, Zatloukal J, Kolek V, Urbanek K, Vasakova M, Stehlik L, Zackova P, Asswad AG. Efficacy and analgesic use during the therapy of iatrogenic pneumothorax using Pleuralvent and Chest Tube (ASPIRATE): A randomised controlled trial protocol. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2020 Jun;164(2):213-215. doi: 10.5507/bp.2020.008. Epub 2020 Mar 9. PMID 32153301